CLINICAL TRIAL: NCT05894252
Title: Walking Interventions to Improve Quality of Life Among Adults with Type 2 Diabetes in Saudi Arabia and the United Kingdom: a Randomised Controlled Trial
Brief Title: Walking Interventions to Improve Quality of Life Among Adults with T2D in SA and the UK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Daniel Lamport, Dr Daniel Lamport, University of Reading
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UReading walking interventions
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Quality of Life
Keywords: Type 2 Diabetes; Intervention; Quality of life; Wellbeing
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: There are 2 groups (i) walking intervention (ii) control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental walking group (Experimental): Participants in the intervention group will need to engage in a 30-minute walk on five days every week for a duration of 12 weeks. To assist them in monitoring their activity and complying with the intervention guidelines, participants will receive a complimentary fitness watch. Weekly step counts will be collected from participants, who will report their data through a researcher-provided online link. The watch will come with an accompanying app for participants to access their data, but the researchers will not have access to this app.
  Interventions: Other: Walking Interventions
- Control (No Intervention): In the control group, participants will not be required to complete the 30 minutes of walking every day. Instead, they will be asked to continue with their daily routines and usual level of physical activity. participants will receive a complimentary fitness watch. Weekly step counts will be collected from participants, who will report their data through a researcher-provided online link. The watch will come with an accompanying app for participants to access their data, but the researchers will not have access to this app.

INTERVENTIONS:
Other: Walking Interventions — Participants in the intervention group will be required to complete a 30-minute walk five days a week for 12 weeks. This will be in addition to any regular walking or exercise they are currently doing, which will be assessed via a questionnaire at baseline. In the control group, participants will be asked to continue with their daily routines and usual level of physical activity.
  The baseline measurements will be taken before the intervention at week zero. Subsequently, all the participants will attend a virtual meeting (screening visit) to learn about the key aspects of the research, including the required actions of the control and intervention groups, how to use the act watch and report the required data. All participants in the intervention group and the control group will be required to wear acti watches, which will be given to them for free.
  Arms: Experimental walking group

SUMMARY:
The research will be conducted as a quantitative experimental study (as an intervention). For the primary DV, quality of life, there are two effective measures.

* Health-related Quality of Life (HRQoL) scales of the SF-36 short form
* Euro-QoL instruments (EQ-5D).

Additionally, secondary variables assessed will be:

* (Physical Activity (the International PA questionnaire, short form - IPAQ)
* General Anxiety (the Generalised Anxiety Disorder Assessment - GAD-7
* Symptoms of Depression (the Patient Health Questionnaire - PHQ-9)
* Habitual diet will be assessed with the EPIC food frequency questionnaire,
* Memory function through the Gorilla online questionnaire (Memory Intrusion - TB1 and TB2).
* Health locus of control (Multidimensional Health Locus of Control form C)

Participants in the intervention group will be required to complete a 30-minute walk five days a week for 12 weeks. This will be in addition to any regular walking or exercise they are currently doing, which will be assessed via questionnaire at baseline. In the control group, participants will be asked to continue with their daily routines and usual level of physical activity.

The baseline measurements will be taken before the intervention at week zero. Subsequently, all the participants will attend a virtual meeting (screening visit) to learn about the key aspects of the research, including the required actions of the control and intervention groups, how to use the act watch and report the required data. All participants in the intervention group and the control group will be required to wear acti-watches, which will be given to them for free.

Participants in both groups will be asked to report the number of steps covered each week. Participants will report this information through an online link provided by the researcher. Each participant will access their data through an app that comes with the watch, however, the researchers will not have access to the app

DETAILED DESCRIPTION:
Diabetes mellitus is a common disease worldwide that affects individuals through physical complications and associated mental health challenges. Physical inactivity among adults with type 2 diabetes is a major public health concern, as it negatively impacts patients' quality of life, especially when they are unable to manage their condition appropriately.

Type 2 diabetes (T2D)-among the leading causes of death and poor quality of life (QoL) in the UK and Saudi Arabia-has two major risk factors: diet and physical activity. The current study will evaluate the efficacy of a walking intervention to improve quality of life of adults with type 2 diabetes in Saudi Arabia and the United Kingdom. A secondary objective is to determine whether the efficacy of the walking intervention differs between populations with type 2 diabetes in the UK and Saudi Arabia.

Participants in the intervention group will be required to complete a 30-minute walk five days a week for 12 weeks. All participants in this study will be required to wear smartwatches or fitness trackers, which will be given to them for free. There will be no direct access to participants' device data for this study; rather, participants will report the data via an online link. Participants, both in the intervention group and in the control group, will be informed of what the study seeks to achieve. In this case, it examines the role of physical activity in health outcomes and quality of life among individuals diagnosed with type 2 diabetes. The experimental group will be given specific instructions to follow for 12 weeks about physical activity. In contrast, the control group will be asked to continue their physical activity as normal for 12 weeks.

The participants will need to have an online screening meeting with the researcher. This will allow the investigator to check whether the participants meet the inclusion criteria. At the screening, participants will complete an online survey that will take approximately 10-15 minutes. The questions will be related to various experiences, physical activity, habitual diet, and feelings associated with diabetes. At the end of the screening session, if participants agree to take part in this study, they will be asked to electronically sign a consent form. Once the screening session is completed, participants will be randomly assigned to one of two groups: the experimental group or the control group.

Assessment will be done via a 30 minute online session at the beginning and end of the 12 week period to measure the following variables: height and weight, blood glucose, physical activity level, anxiety, depression, quality of life, and memory function. A fitness tracker acti-watch will be used to track the physical activity of participants. This will be provided to participants free of charge. Participants will be asked to report their total number of steps each week via an online link provided by the researcher on a weekly basis.

Two versions of all research materials will be created (English and Arabic). To ensure reliability, all the Arabic versions of the questionnaires have been independently validated and published elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes.
* Residing in the UK or Saudi Arabia.
* Must have access to the internet once a week to answer questions via an online link.
* Adults (18 - 64 years)

Exclusion Criteria:

* Being unable to walk.
* Pregnant or given birth in the last 12 months
* Scoring a high levels of physical activity on the international physical activity questionnaire - short form. An individual with more than 3000 MET minutes a week will be considered to have a high level of PA according to the survey authors

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Quality of life (EQ-5D-5L) t1 | Baseline week zero
  The five-dimensional EuroQol scale will be used to assess the quality of life (EQ-5D-5L). The EQ-5D-5L is based on a descriptive system that consists of five dimensions, each capturing a different aspect of health-related quality of life. These dimensions are mobility, self-care, usual activities pain/discomfort, and anxiety/depression each dimension is rated on a five-level scale, which allows individuals to indicate their level of problems or impairment. The five levels are no problems, slight problems, moderate problems, severe problems, and extreme problems. The combination of responses creates a unique health state profile, which can be converted into a single index value representing overall health status. This index value ranges from 0 (representing the worst possible health state) to 1 (representing full health). Higher scores indicate a higher level of health-related quality of life.
Quality of life (EQ-5D-5L) t2 | Week 12
  The five-dimensional EuroQol scale will be used to assess the quality of life (EQ-5D-5L). The EQ-5D-5L is based on a descriptive system that consists of five dimensions, each capturing a different aspect of health-related quality of life. These dimensions are mobility, self-care, usual activities pain/discomfort, and anxiety/depression each dimension is rated on a five-level scale, which allows individuals to indicate their level of problems or impairment. The five levels are no problems, slight problems, moderate problems, severe problems, and extreme problems. The combination of responses creates a unique health state profile, which can be converted into a single index value representing overall health status. This index value ranges from 0 (representing the worst possible health state) to 1 (representing full health). Higher scores indicate a higher level of health-related quality of life.
Quality of life Short Form 36 Health Survey Questionnaire (SF-36) t1 | Baseline week zero
  A second measure of quality of life will be obtained by completing the Short Form 36 Health Survey Questionnaire (SF-36).The Short Form 36 Health Survey Questionnaire (SF-36) is a used as self-reported instrument assessing health-related quality of life (HRQoL). It consists of 36 questions measuring physical and mental health across eight dimensions. Physical health includes functioning, role limitations, pain, and general health perceptions. Mental health covers vitality, social functioning, role limitations, and mental health. Each dimension is scored from 0 to 100, with higher scores indicating better HRQoL.
Quality of life Short Form 36 Health Survey Questionnaire (SF-36) t2 | Week 12
  A second measure of quality of life will be obtained by completing the Short Form 36 Health Survey Questionnaire (SF-36). The Short Form 36 Health Survey Questionnaire (SF-36) is a used as self-reported instrument assessing health-related quality of life (HRQoL). It consists of 36 questions measuring physical and mental health across eight dimensions. Physical health includes functioning, role limitations, pain, and general health perceptions. Mental health covers vitality, social functioning, role limitations, and mental health. Each dimension is scored from 0 to 100, with higher scores indicating better HRQoL.

SECONDARY OUTCOMES:
Anxiety t1 | Baseline week zero
  The Generalized Anxiety Disorder 7-item scale (GAD-7) is a self-report questionnaire designed to assess the severity of generalized anxiety disorder symptoms. It consists of seven questions that capture common anxiety symptoms experienced over the past two weeks. Individuals rate the frequency of symptoms on a scale from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 21, with higher scores indicating greater anxiety severity.
Anxiety t2 | Week 12
  The Generalized Anxiety Disorder 7-item scale (GAD-7) is a self-report questionnaire designed to assess the severity of generalized anxiety disorder symptoms. It consists of seven questions that capture common anxiety symptoms experienced over the past two weeks. Individuals rate the frequency of symptoms on a scale from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 21, with higher scores indicating greater anxiety severity.
Depression t1 | Baseline week zero
  An assessment of depression symptoms is conducted with the Patient Health Questionnaire 9-item scale (PHQ-9). It consists of nine questions that capture common depressive symptoms experienced over the past two weeks. Each item is rated on a scale from 0 (not at all) to 3 (nearly every day), reflecting the frequency and intensity of symptoms. The total score ranges from 0 to 27, with higher scores indicating greater depression severity.
Depression t2 | Week 12
  An assessment of depression symptoms is conducted with the Patient Health Questionnaire 9-item scale (PHQ-9). It consists of nine questions that capture common depressive symptoms experienced over the past two weeks. Each item is rated on a scale from 0 (not at all) to 3 (nearly every day), reflecting the frequency and intensity of symptoms. The total score ranges from 0 to 27, with higher scores indicating greater depression severity.
Exercise level (The International Physical Activity Questionnaires) (IPAQ) t1 | Baseline week zero
  Physical activity levels are assessed using the International Physical Activity Questionnaires (IPAQ). A number of versions of the IPAQ are available, including the IPAQ-LF (long form) and IPAQ-SF (short form). The IPAQ-LF collects detailed information about work, transportation, chores, and leisure activities and provides an estimate of total physical activity. IPAQ-SF focuses on walking, moderate, and vigorous activities, giving domain-specific and total estimates. This study will use a short-form version of the IPAQ (IPAQ-SF). The total score for IPAQ varies based on reported activity levels across domains. It can range from 0 (no activity) to higher values indicating significant weekly physical activity.
Exercise level (The International Physical Activity Questionnaires) (IPAQ) t2 | Week 12
  Physical activity levels are assessed using the International Physical Activity Questionnaires (IPAQ). A number of versions of the IPAQ are available, including the IPAQ-LF (long form) and IPAQ-SF (short form). The IPAQ-LF collects detailed information about work, transportation, chores, and leisure activities and provides an estimate of total physical activity. IPAQ-SF focuses on walking, moderate, and vigorous activities, giving domain-specific and total estimates. This study will use a short-form version of the IPAQ (IPAQ-SF). The total score for IPAQ varies based on reported activity levels across domains. It can range from 0 (no activity) to higher values indicating significant weekly physical activity.
Food frequency Epic FFQ t1 | Baseline week zero
  Food Frequency Epic FFQ is a questionnaire that assesses dietary intake. It collects data on food frequency and portion sizes, estimating nutrient and food group intakes. Participants report average consumption over a defined period.
Food frequency Epic FFQ t2 | Week 12
  Food Frequency Epic FFQ is a questionnaire that assesses dietary intake. It collects data on food frequency and portion sizes, estimating nutrient and food group intakes. Participants report average consumption over a defined period.
Cognitive functionality (Memory) t1 | Baseline week zero
  The Memory Intrusion - TB1&TB2 paradigm is a widely used method to study memory retrieval and false memory effects. Participants memorize a list of words and then indicate if words in a second list were present in the original (old) or not (new). The second list includes related foils, leading to false memories. This paradigm sheds light on memory processes and factors affecting accuracy in cognitive.
Cognitive functionality (Memory) t2 | Week 12
  The Memory Intrusion - TB1&TB2 paradigm is a widely used method to study memory retrieval and false memory effects. Participants memorize a list of words and then indicate if words in a second list were present in the original (old) or not (new). The second list includes related foils, leading to false memories. This paradigm sheds light on memory processes and factors affecting accuracy in cognitive.
Steps Smartwatch | Repeated weekly. Week 1
  Participants are required to log in to a link once a week and self-report their total steps for the week. This simple process allows for regular tracking of participants' physical activity levels, promoting engagement and accountability in monitoring their step counts.
Steps Smartwatch | Repeated weekly. Week 2
  Participants are required to log in to a link once a week and self-report their total steps for the week. This simple process allows for regular tracking of participants' physical activity levels, promoting engagement and accountability in monitoring their step counts.
Steps Smartwatch | Repeated weekly. Week 3
  Participants are required to log in to a link once a week and self-report their total steps for the week. This simple process allows for regular tracking of participants' physical activity levels, promoting engagement and accountability in monitoring their step counts.
Steps Smartwatch | Repeated weekly. Week 4
  Participants are required to log in to a link once a week and self-report their total steps for the week. This simple process allows for regular tracking of participants' physical activity levels, promoting engagement and accountability in monitoring their step counts.
Steps Smartwatch | Repeated weekly. Week 5
  Participants are required to log in to a link once a week and self-report their total steps for the week. This simple process allows for regular tracking of participants' physical activity levels, promoting engagement and accountability in monitoring their step counts.
Steps Smartwatch | Repeated weekly. Week 6
  Participants are required to log in to a link once a week and self-report their total steps for the week. This simple process allows for regular tracking of participants' physical activity levels, promoting engagement and accountability in monitoring their step counts.
Steps Smartwatch | Repeated weekly. Week 7
  Participants are required to log in to a link once a week and self-report their total steps for the week. This simple process allows for regular tracking of participants' physical activity levels, promoting engagement and accountability in monitoring their step counts.
Steps Smartwatch | Repeated weekly. Week 8
  Participants are required to log in to a link once a week and self-report their total steps for the week. This simple process allows for regular tracking of participants' physical activity levels, promoting engagement and accountability in monitoring their step counts.
Steps Smartwatch | Repeated weekly. Week 9
  Participants are required to log in to a link once a week and self-report their total steps for the week. This simple process allows for regular tracking of participants' physical activity levels, promoting engagement and accountability in monitoring their step counts.
Steps Smartwatch | Repeated weekly. Week 10
  Participants are required to log in to a link once a week and self-report their total steps for the week. This simple process allows for regular tracking of participants' physical activity levels, promoting engagement and accountability in monitoring their step counts.
Steps Smartwatch | Repeated weekly. Week 11
  Participants are required to log in to a link once a week and self-report their total steps for the week. This simple process allows for regular tracking of participants' physical activity levels, promoting engagement and accountability in monitoring their step counts.
Steps Smartwatch | Repeated weekly. Week 12
  Participants are required to log in to a link once a week and self-report their total steps for the week. This simple process allows for regular tracking of participants' physical activity levels, promoting engagement and accountability in monitoring their step counts.
Health Locus Control (Multidimensional Health Locus of Control form C- MHLC) t1 | Baseline week zero
  The MHLC-C assesses health control beliefs for individuals with a medical condition across four subscales: Internal, Chance, Doctors, and Others. Scores range from 6 to 36 per subscale, and the overall score spans 18 to 108. Higher Internal scores indicate increased belief in personal control over health outcomes. Elevated scores on Chance, Doctors, and Others suggest reliance on external factors, with varied interpretations. A higher Doctors score may imply trust in medical professionals, while raised Chance or Others scores may indicate a perceived lack of personal control. Overall, higher MHLC-C scores denote a more external health locus of control, attributing health outcomes to factors beyond personal control.
Health Locus Control (Multidimensional Health Locus of Control form C- MHLC) t2 | Week 12
  The MHLC-C assesses health control beliefs for individuals with a medical condition across four subscales: Internal, Chance, Doctors, and Others. Scores range from 6 to 36 per subscale, and the overall score spans 18 to 108. Higher Internal scores indicate increased belief in personal control over health outcomes. Elevated scores on Chance, Doctors, and Others suggest reliance on external factors, with varied interpretations. A higher Doctors score may imply trust in medical professionals, while raised Chance or Others scores may indicate a perceived lack of personal control. Overall, higher MHLC-C scores denote a more external health locus of control, attributing health outcomes to factors beyond personal control.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lamport, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom